CLINICAL TRIAL: NCT07360938
Title: Drug Interaction Potential of Pro-Inflammatory Conditions
Acronym: DIPPIC
Status: Recruiting | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Tyler Andrew Shugg, Assistant Professor, Indiana University
Other Study IDs: 27983
Record Dates: First submitted 2026-01-06; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 2; End Stage Renal Disease; Irritable Bowel Syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Kidney Failure, Chronic; Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Type 2 Diabetes Mellitus
  Interventions: Other: None (Observational)
- End Stage Renal Disease
  Interventions: Other: None (Observational)
- Irritable Bowel Syndrome
  Interventions: Other: None (Observational)

INTERVENTIONS:
Other: None (Observational) — This observational study will not involve any interventions. Instead, the study will collect blood samples at one or multiple time points.

SUMMARY:
Pro-inflammatory cytokines, which are elevated in pro-inflammatory disease states (e.g., type II diabetes mellitus [T2DM], irritable bowel diseases [IBD], and end stage renal disease [ESRD]) have been shown to inhibit hepatic drug-metabolizing enzymes, including members of the cytochrome P450 (CYP) family, and drug transporters; resultantly, pro-inflammatory diseases have been demonstrated to increase the exposure and potential for adverse drug events with co-administered CYP and drug transporter substrates. However, the clinical relevance of pro-inflammatory disease-drug interactions has not been systematically evaluated. The long-term goal of this research is to establish clinical strategies to mitigate pro-inflammatory disease-drug interactions and associated adverse drug events. The specific objective of this study is to determine the clinical relevance of pro-inflammatory disease-drug interactions, including establishment of the effect of pro-inflammatory diseases on drug disposition throughout disease trajectories (i.e., determining the differential effects on drug disposition based on the severity of disease). Towards this objective, this study will investigate the extent of increases in inflammation in patients with varying severities of pro-inflammatory diseases and estimate the resulting effects on drug disposition. Cytokine/chemokine concentrations and immune cell profiles will be assayed from blood samples of adult and pediatric patients with differing severities of pro-inflammatory diseases, using established disease monitoring parameters (e.g., glycosylated hemoglobin [HbA1C] for T2DM, C-reactive protein [CRP] for IBD, proteinuria for ESRD). The effect of changes in inflammation during differing severities of these pro-inflammatory diseases on drug disposition will then be estimated using established pharmacokinetic modeling approaches (e.g., physiologically-based pharmacokinetic modeling [PBPK]).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a pro-inflammatory disease, including T2DM, IBD, and ESRD
* Ability to provide written informed consent and HIPAA authorization

Exclusion Criteria:

* Diagnosis or past medical history of non-IBD autoimmune disorder, including systemic lupus erythematosus, Sjogren's syndrome, multiple sclerosis, type 1 diabetes mellitus, Behcet's disease, and ankylosing spondylitis
* Current infection requiring medical treatment (note: if a prospective patient's infection resolves, they can be re-screened for trial inclusion)
* Concomitant treatment with systemic immunosuppressant drugs

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a prospective observational study that will collect blood samples at 1-3 timepoints per patient. The study will not include any therapeutic intervention, and no study visits will involve patient interaction with the health system solely for study participation. The study will enroll up to 150 patients. All enrolled patients will undergo the study procedures, which will enable quantification of plasma cytokine concentrations and immune cell profiles at 1-3 timepoints.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantification of Plasma Cytokine Concentrations | Through study completion, up to 2 years post enrollment
  The first primary objective will involve quantification of plasma cytokine concentrations from patient blood samples.
Phenotyping of Patient Immune Cells | Through study completion, up to 2 years post enrollment
  The second primary objective will involve phenotyping of patient immune cells from patient blood samples.
Quantification of the Plasma Concentrations of Endogenous Biomarkers of Drug Metabolism and Transport | Through study completion, up to 2 years post enrollment
  The third primary objective will involve quantification of the plasma concentrations of endogenous biomarkers of drug metabolism and transport from patient blood samples
Measures of Inflammatory Disease Severity | Through study completion, up to 2 years post enrollment
  The fourth primary objective will involve collecting measures of inflammatory disease severity based on information collected from patients' electronic health records.
Development of Adverse Events Attributable to CYP/Transporter Substrate Medications | Through study completion, up to 2 years post enrollment
  The fifth primary objective will involve collecting the development of adverse drug events attributable to CYP/transporter substrate medications based on information collected from patients' electronic health records.

SECONDARY OUTCOMES:
Patient Genomic Markers | Through study completion, up to 2 years post enrollment
  The secondary objective will involve determining patient genomic markers (using whole genome sequencing).

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
There are Material Transfer Agreements and Data Use Agreements in place to share IPD.